CLINICAL TRIAL: NCT04212351
Title: Frameshift Peptides of Children With Neurofibromatosis Type 1 (NF1) and Either Low-Grade Gliomas or Plexiform Neurofibromas
Brief Title: Frameshift Peptides of Children With NF1
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Arizona State University (Other); Emory University (Other)
Responsible Party: Principal Investigator, Roger Packer, Senior Vice President of Neurology and Behavorial Medicine, Children's National Research Institute
Other Study IDs: Pro00011544
Record Dates: First submitted 2019-05-01; First posted 2019-12-27 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A frameshift peptide profile will be determined from patient blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with NF1 and active LGGs: Patients with Neurofibromatosis Type 1 with clinical or radiographic evidence of low grade glioma but no clinical or radiographic evidence of plexiform neurofibroma.
  Interventions: Genetic: Frameshift Array blood sample test
- Patients with NF1 and active PNs: Patients with Neurofibromatosis Type 1 with clinical or radiographic evidence of plexiform neurofibroma but no clinical or radiographic evidence of low grade glioma.
  Interventions: Genetic: Frameshift Array blood sample test
- Patients with NF1 with no active LGGs or PNs: Patients with Neurofibromatosis Type 1 with no clinical or radiographic evidence of both active plexiform neurofibroma and active low grade glioma.
  Interventions: Genetic: Frameshift Array blood sample test

INTERVENTIONS:
Genetic: Frameshift Array blood sample test — Patient blood test samples will be collected and evaluated for frameshift peptide mutations.

SUMMARY:
The objective of this study is to determine if children and young adults with Neurofibromatosis Type 1 (NF1) and either Low Grade Gliomas (LGGs) or Plexiform Neurofibromas (PNs) have a specific frameshift peptide protein profile and whether a disease specific vaccine created to address these frameshift mutations and variants can be developed. Three study populations will be analyzed; patients with NF1 and active LGGs, NF1 and active PNs, and NF1 and no evidence of active LGGs or PNs. Participation involves a onetime blood draw.

DETAILED DESCRIPTION:
I. Objective and Specific Aims

A. Objectives:

To determine if children and young adults with NF1 and either Low Grade Gliomas (LGGs) or Plexiform Neurofibromas (PNs) have a specific frameshift peptide protein profile and whether a disease specific vaccine created to address these frameshift mutations and variants can be developed.

B. Primary Aims:

1. Determine the frameshift peptide profile of children and young adults with NF1 and active LGGs, NF1 and active PNs, and NF1 and no evidence of active LGGs or PNs.
2. Determine if the frameshift peptide profiles of children and young adults with NF1 in each of the populations of interest differ.
3. Determine if specific frameshift peptide profiles can be used to create a disease specific vaccine for children and young adults with NF1 and either LGGs or PNs.

C. Secondary Aims:

1. To assess the impact of age, gender, family history of NF, disease state (stable, progressive, or responding), and treatment on the frameshift peptide profiles of children and young adults with NF1 and active LGGs or PNs.
2. To assess the impact of NF1 mutation type on the frameshift peptide profiles found.

II. Background

A. Neurofibromatosis Type 1

Neurofibromatosis Type I (NF1) is a genetic disorder that affects 1 in 3000 individuals caused by a germline heterozygous mutation of the NF1 gene located on chromosome 17. Inherited as an autosomal dominant gene, the mutation is 100% penetrant and is manifested by multiple complications, many of which can significantly inhibit an individual's ability to function in daily life and, in some cases, may be life threatening (Viskochil et al., 1990, Wallace et al., 1990). To date, only a variable association has been made between the type of mutation present and the phenotype of the affected individual. Some manifestations of NF1, such as café au lait spots and dermal fibromas, are extremely common while others, although less frequent, may cause severe neurologic or other organ dysfunction (Ferner et al., 2007). Two of the most common NF1-related manifestations are plexiform neurofibromas and gliomas, especially gliomas affecting the visual system. Treatment for both is currently suboptimal, however new molecularly targeted and immunologic approaches hold the promise of improved outcomes (Khatua et al., 2018).

Gliomas may develop as early as infancy with an initial peak in diagnosis between the ages of 3 and 5 years (Schmandt & Packer, 2000, Khatua et al., 2018). At the time of clinical detection, there is often significant tumor associated morbidity frequently resulting in irreversible visual impairment, which may worsen as these tumors of the optic nerve and chiasm progress. Therapies are currently available to slow or stop the growth of these lesions; however, these therapies often do not halt visual loss, rarely result in visual improvement, and may only be of transient benefit. Gliomas may also arise in different areas of the brain, especially in the brain stem later in childhood and into early adulthood. When these tumors become active in adolescents or young adults, they may mutate into more aggressive anaplastic pilocytic astrocytomas and become resistant to therapy. These more aggressive gliomas are a potential cause of death in patients with NF1.

Plexiform neurofibromas may occur in up to 60% of NF1 patients with the potential to result in severe disfigurement and neurologic compromise by compression of the spinal cord or peripheral nerves (Packer et al., 2018). Depending on location, plexiform neurofibromas may also result in severe respiratory compromise or urologic dysfunction. Although believed to be congenital manifestations, many may not become evident or symptomatic until later in life. Between 6-13% of plexiform neurofibromas will mutate into malignant peripheral nerve sheath lesions, which typically respond poorly to current therapeutic options and can result in death.

Patients with NF1 have a shortened life expectancy compared to those without due, in part, to the devastating plexiform neurofibromas, malignant peripheral nerve sheath tumors, and gliomas they develop (Packer et al., 2018). A clinically important question in NF1 patients is whether the diagnosis and treatment of incipient tumors will result in better outcomes and decrease the likelihood of malignant progression of those tumors. Recent advances in imaging and image processing have improved the precision and detail of visualization of the growing tumor mass, however, it would be ideal to develop a blood test capable of indicating the status of these NF1 children. Early interventions with better treatments may prove more effective and less harmful to the patient than more aggressive treatments needed at a later stage of disease. Furthermore, treatment by immunotherapeutic approaches, especially the development of a vaccine to prevent the occurrence or progression of gliomas and plexiform neurofibromas, is a potentially function saving and lifesaving intervention.

III. Methods

Each enrolled participant will undergo a one-time blood draw, collecting up to 10ml. Study sites will also obtain basic demographic and clinical information.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 1 day and 30 years of age, inclusive
2. Subjects must either meet clinical criteria for NF1 or have molecular genetic germ line evidence of NF1
3. Subject is able to have his/her blood sample drawn within a reasonable period of time after signing consent
4. Subjects must either have:

   1. Active* LGGs, no active PNs (Cohort 1)
   2. Active* PNs, no active LGGs (Cohort 2)
   3. No active* LGGs or PNs (Cohort 3) *Active is defined as any LGG or PN that has shown growth (determined by MRI) in the past 12 months or is causing ongoing symptomatic visual, neurologic, or organ dysfunction or disfigurement as determined by the site investigator.

Exclusion Criteria:

1. Patients with NF1 with evidence of both LGG and PN

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: There will be a total of 60 patients enrolled in the study. Cohort 1 will consist of 20 subjects with NF1 and active LGG. Cohort 2 will consist of 20 subjects with NF1 and active PN. Cohort 3 will consist of 20 subjects with NF1 and no active LGG or active PN.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Measure mean florescent intensity of serum/plasma samples for each cohort by assaying the study samples on frameshift peptide arrays consisting of peptides representing the ~220,000 frameshifts tumors can make in RNA processing. | 2 years
  All samples will be assayed on the FSP arrays consisting of peptides representing the frameshifts tumors can make in RNA processing. The amount of IgG bound to each feature will be determined as florescent intensity generated by bound secondary antibody. The mean intensity across the 20 subjects for each peptide for each of the 3 groups will be determined. All peptides in the NF1+LGG group with mean intensities greater than 3 SD higher than the mean of the NF1-LGG/PN group will be determined. Those that meet this criterion in more than 3 of the 20 samples will be chosen. The 20 peptides with the highest prevalence across the 20 samples of NF1+LGG will be chosen for the vaccine. If two peptides have the same prevalence, the one with the highest average florescence will be chosen. The same procedure will be applied to determine the 20 peptide components for the NF1+PN vaccine.
Use a feature counting method to establish a mean distinguishable frameshift peptide protein profile for early detection of tumors in patients with NF1. | 2 years
  The same data as generated in Outcome 1 will be analyzed for the ability to distinguish NF1+LGG and NF1+PN samples from the NF1-LGG/PN samples. Since the antibody reactions to frameshift peptides are stochastic, a feature counting method is employed. A mean is established for each of the NF1-LGG/PN peptides. Any peptide in the NF1+LGG and NF1+PN samples that scores 3 SD higher than NF1-LGG/PN mean is scored as a positive. The total number of positives in the NF1+LGG and NF1+PN pool will be compared to that in the NF1-LGG/PN set. The number of samples that are distinguished by these counts will determine a first pass accuracy estimate of this diagnostic approach as a preamble to an expanded study.
Use a feature counting method to establish a mean distinguishable frameshift peptide protein profile for patient who develop LGGs versus patients who develop PNs. | 2 years
  The same array data generated in Outcome 1 will be used. The feature counting method used in Outcome 2 will be used to compare the NF1+LGG features to the NF1+PN features. The investigators will determine if there are a set of features that can distinguish the 20 NF1+LGG from the 20 NF1+PN samples. The number of NF1+LGG and NF1+PN samples that can be distinguished will provide a first estimate of accuracy and whether an expanded study is merited.

SECONDARY OUTCOMES:
Correlate age, gender, family history of NF, disease state (stable, progressive, or improving), and disease history with frameshift peptide profiles, in children and young adults with NF1 and LGGs or PNs. | 2 years
  Correlate age, gender, family history of NF, disease state (stable, progressive, or improving), and disease history with frameshift peptide profiles, in children and young adults with NF1 and LGGs or PNs.

CONTACTS AND LOCATIONS:
Overall Officials: Roger J. Packer, MD, Principal Investigator — Children's National Research Institute
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - The University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers outside of Children's National Medical Center.